CLINICAL TRIAL: NCT00803387
Title: Dry Eye and Irritation Comparison of Latanoprost 0.005% With the Preservative Benzalkonium Chloride (BAC) Vs Travoprost 0.004% Without BAC
Brief Title: Dry Eye and Irritation Comparison of Latanoprost With the Preservative Versus Travoprost Without Preservative
Status: Completed | Type: Observational
Sponsor: United States Air Force (U.S. Federal Agency)
Collaborators: Alcon Research (Industry)
Responsible Party: Capt James Richard Townley, MD, USAF
Other Study IDs: FWH20080020H
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2008-12-05 (Estimated); Status verified 2008-12

CONDITIONS: Ocular Dryness; Ocular Irritation; Open-Angle Glaucoma; Ocular Hypertension
Keywords: ocular dryness; ocular irritation; open-angle glaucoma; ocular hypertension; TravatanZ; Xalatan
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Bacitracin; Travoprost

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients taking Xalatan with ocular dryness or irritation: * patient must already be using xalatan for at least 1 month prior to study enrollment in both eyes and have complaints of dry eye and/or irritation.
  * any race and of either sex, diagnosed with open angle glaucoma (OAG) (with or without pseudoexfoliation or pigment dispersion components) or ocular hypertension (OHT)
  Interventions: Drug: Travaprost without BAC (Travatan Z)

INTERVENTIONS:
Drug: Travaprost without BAC (Travatan Z) — A double blind comparison was used to assess whether Xalatan or TrvatanZ affects the tear breakup times, corneal staining, and baseline tear secretion tests in patients that are already taking latanoprost regularly with complaints of dryness and irritation. Patients included in the study will be given two bottles, one labeled for their right eye and the other for their left eye. Each pair of bottles will be identical in appearance and randomized with either latanoprost or travoprost and each pair will be assigned a number to aid in future analysis of the final results. One Drop from both bottles will be dispensed in the respective eye once a day.

SUMMARY:
Although Benzalkonium chloride (BAC) has been used as a preservative for many years, many studies have demonstrated that prolonged use of topical ocular medications preserved with BAC may exacerbate sequelae associated with ocular surface disease. These effects could lead to the induction of subclinical inflammation,1 reduction of corneal epithelial barrier function, 2, 3 destabilization of the tear film, 4 cataract formation, 5 and an overall higher incidence of patient complaints of dryness and irritation. 4-6 This study will compare the efficacy of travoprost 0.004% without benzalkonium chloride (BAC) to that of the marketed formulation of latanoprost 0.005%with BAC in patients with dryness and irritation and open-angle glaucoma or ocular hypertension. A double blind comparison will be used to assess whether those two different formulations will affect the tear breakup times, corneal staining, and baseline tear secretion tests in patients that are already taking latanoprost regularly with complaints of dryness and irritation. Patients included in the study will be given two bottles, one labeled for their right eye and the other for their left eye. Each pair of bottles will be identical in appearance and randomized with either latanoprost or travoprost and each pair will be assigned a number to aid in future analysis of the final results.

ELIGIBILITY:
Inclusion Criteria:

* patient must already be using xalatan for at least 1 month prior to study enrollment in both eyes and have complaints of dry eye and/or irritation.
* study population:
* any race and of either sex, diagnosed with open angle glaucoma (OAG) (with or without pseudoexfoliation or pigment dispersion components) or ocular hypertension (OHT)
* tear break up times (TBUT) < 6 seconds on xalatan monotherapy.

Exclusion Criteria:

* unequal baseline measurements (i.e. difference in cup to disc ratio of .1 or greater, intraocular pressure difference of 2 or more mm Hg),
* difference in subjective symptoms of dryness/irritation between the patient's two eyes;
* history of ocular trauma or intraocular surgery within the past 6 months in either eye;
* ocular infection, ocular inflammation, or ocular laser surgery within the past 3 months in either eye;
* severe hypersensitivity to study medications or vehicle;
* any abnormality preventing reliable applanation tonometry;
* anterior chamber angle less than 10 degrees in either eye,
* severe central visual field loss in either eye;
* cup-to-disc ratio greater than 0.80 in either eye;
* contraindications to pupil dilation; previous diagnosis of autoimmune diseases;
* chronic glucocorticoid use within 1 month of and during the eligibility phase or intermittent glucocorticoid use within 2 weeks of the eligibility phase;
* any type of glaucoma other than OAG or OHT;
* therapy with another investigational agent within 30 days of study start;
* use of any other topical or systemic ocular hypotensive medication during the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Must be eligible for care at WHMC ie active duty, military retirees and their dependents
  * patient must already be using xalatan for at least 1 month prior to study enrollment in both eyes and have complaints of dry eye and/or irritation.
  * any race and of either sex, diagnosed with open angle glaucoma (OAG) (with or without pseudoexfoliation or pigment dispersion components) or ocular hypertension (OHT)
  * tear break up times (TBUT) < 6 seconds on xalatan monotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2008-04; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Routine eye exams in addition to Ocular Surface Disease Index (OSDI) surveys at the beginning and end of the study. Patients will also be asked to rate their extent of dryness and irritation of either eye on a scale of 1-10 at each visit. | Each patient will be followed every 3-4 weeks for 3 months

CONTACTS AND LOCATIONS:
Overall Officials: James R Townley, MD, Principal Investigator — United States Air Force
Locations (1):
- WHMC, Lackland Air Force Base, Texas, United States